CLINICAL TRIAL: NCT01052597
Title: Antiatherogenic and Antimetabolic Effect of Curcumin in Type 2 Diabetic Patients
Brief Title: Curcumin for Type 2 Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Srinakharinwirot University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Assist.Prof. Somlak Chuengsamarn, Department of Internal Medicines, Faculty of Medicine, Srinakarinwirot University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWUEC30/2550
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2007-08

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Abnormalities
Keywords: Type 2 diabetes; Metabolic syndrome; cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Abnormalities; Metabolic Syndrome | interventions — Curcumin; Tacrine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: curcumin
- Curcumin (Experimental)
  Interventions: Drug: curcumin

INTERVENTIONS:
Drug: curcumin — Curcumin capsule contains 250 mg curcuminoids, 2 capsule per time, 3 times a day for 12 months
  Other Names: Manufactured by Government Pharmaceutical Organization, Thailand

SUMMARY:
There are evidence that there is an association between insulin resistance and prolonged hyperinsulinemia or hyperglycemia in Type 2 diabetic patients. This will trigger oxidative stress system via reactive oxygen species (ROS) and lead to a high level of Nitric oxide. This can contribute to a significant change in blood vessel and could end up with the complications from cardiovascular disease and increased mortality rate of type 2 diabetic patients. The purpose of the present study was to examine the effectiveness of the curcumin in type 2 diabetic patients on the reduction of atherosclerosis events by examining pulse-wave velocity (PWV) and plasma high-sensitivity C-reactive protein (CRP) test and on blood sugar lowering, glycosylated hemoglobin (HBA1c), lipid profile, and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients aged 35 years or older and did not use insulin during the first 5 years of treatment after being diagnosed (with or without symptoms listed in the following inclusion criteria)
* Patient with hyperlipidemia (Cholesterol ≥ 200 mg/dl, TG ≥ 150 mg/dl, LDL ≥ 100 mg/dl and HDL ≥ 35 mg/dl)
* Patient with hypertension (Blood pressure ≥ 130/85 mmHg or take hypertensive drugs)
* Obesity (BMI ≥ 25)

Exclusion Criteria:

* Current diagnosis of secondary peripheral arterial disease (PAD) (except listed in the inclusion criteria item 1-4)
* Current diagnosis of cardiovascular disease, i.e., coronary arterial disease and cerebrovascular disease
* Current diagnosis of end stage renal function with serum creatinine > 2.0 mg/dl or on renal dialysis
* Current diagnosis of cirrhosis with ALT ≥ 3 times of normal range

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
to determine the effectiveness of curcumin on reduction of atherosclerotic events and risks in Type 2 diabetic patients | 12 months

SECONDARY OUTCOMES:
To examine the effectiveness of curcumin on the reduction of blood sugar, glycosylated hemoglobin (HBA1c), lipid profile, and insulin resistance | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Somlak Chuengsamarn, Medical Doctor, Principal Investigator — Srinakarinwirot University
Locations (1):
- HRH Princess Maha Chakri Sirindhorn Medical Center, Ongkarak, Nakornnayok, Thailand

REFERENCES:
- [Derived] Chuengsamarn S, Rattanamongkolgul S, Phonrat B, Tungtrongchitr R, Jirawatnotai S. Reduction of atherogenic risk in patients with type 2 diabetes by curcuminoid extract: a randomized controlled trial. J Nutr Biochem. 2014 Feb;25(2):144-50. doi: 10.1016/j.jnutbio.2013.09.013. Epub 2013 Nov 6. PMID 24445038